CLINICAL TRIAL: NCT01122940
Title: Bioequivalence Study Of 10ml Dose Of Phenytoin 0.75g/100ml Suspension Made By Laboratorios Pfizer, S.A. De C.V. Versus Epamin® 0.75g/100ml Made By McNeil LA LLC, Study In 34 Healthy Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study Of Phenytoin Suspension Versus Epamin® In 34 Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A4121008
Record Dates: First submitted 2010-04-20; First posted 2010-05-13 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2011-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Phenytoin; Epamin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epamin: McNeil LA LLC (Active Comparator)
  Interventions: Drug: Epamin: Reference Drug
- Phenytoin: Laboratorios Pfizer SA DE CV (Experimental)
  Interventions: Drug: Phenytoin: Study Drug

INTERVENTIONS:
Drug: Epamin: Reference Drug — Single dose of 75 mg (10 ml in suspension) of Epamin
  Arms: Epamin: McNeil LA LLC
Drug: Phenytoin: Study Drug — Single dose of 75 mg (10 ml in suspension) of Phenytoin
  Arms: Phenytoin: Laboratorios Pfizer SA DE CV

SUMMARY:
Mexican healthy volunteers will receive the current form of the drug (under the name of Epamin) as well as Pfizer's compound (Phenytoin). Bioequivalence will be tested.

DETAILED DESCRIPTION:
Bioequivalence

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive
* A Body Mass Index (BMI) of 18 to 26.9 kg/m2 or ± 10% variation of the ideal weight; and a total body weight >50 kg (110 lbs)
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Any condition possibly affecting drug absorption (eg, gastrectomy)
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To prove the bioequivalence of Phenytoin versus Epamin by measuring; Area under the curve (AUC), Maximum Concentration (Cmax), Time maximum concentration (tmax), Constant of elimination (ke), Elimination half life (t1/2) | April 2010 - May 2010

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4121008&StudyName=Bioequivalence%20Study%20Of%20Phenytoin%20Suspension%20Versus%20Epamin%AE%20In%2034%20Healthy%20Volunteers.